CLINICAL TRIAL: NCT00117312
Title: An Open-Label, Multi-Center, Extension Study Investigating the Long-Term Safety and Tolerability of Repeat Doses of FE200486 in Prostate Cancer Patients
Brief Title: Extension Study Investigating the Long-Term Safety and Tolerability of Repeat Doses of FE200486 in Prostate Cancer Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: After 190 weeks [7 patients left] it was terminated for administrative reasons
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Clinical Development Support, Ferring Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FE200486 CS06A
Record Dates: First submitted 2005-06-30; First posted 2005-07-06 (Estimated); Results first posted 2009-03-20 (Estimated); Last update posted 2011-05-23 (Estimated); Status verified 2011-05

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Androgen ablation therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Degarelix 40 mg (Experimental): Degarelix 40 mg (10 mg/mL)
  Interventions: Drug: Degarelix
- Degarelix 80 mg (Experimental): Degarelix 80 mg (20 mg/mL)
  Interventions: Drug: Degarelix
- Degarelix 120 mg (Experimental): Degarelix 120 mg (30 mg/mL)
  Interventions: Drug: Degarelix
- Degarelix 160 mg (Experimental): Degarelix 160 mg (40 mg/mL)
  Interventions: Drug: Degarelix

INTERVENTIONS:
Drug: Degarelix — One dose (2 x 2 mL) of degarelix 40 mg (10 mg/mL), subcutaneous injection.
  Other Names: FE200486
  Arms: Degarelix 40 mg
Drug: Degarelix — One dose (2 x 2 mL) of degarelix 80 mg (20 mg/mL), subcutaneous injection.
  Other Names: FE200486
  Arms: Degarelix 80 mg
Drug: Degarelix — One dose (2 x 2 mL) of degarelix 120 mg (30 mg/mL), subcutaneous injection.
  Other Names: FE200486
  Arms: Degarelix 120 mg
Drug: Degarelix — One dose (2 x 2 mL) of degarelix 160 mg (40 mg/mL), subcutaneous injection.
  Other Names: FE200486
  Arms: Degarelix 160 mg

SUMMARY:
Participants responding well in Study FE200486 CS06 (NCT00117949) were given the opportunity to continue treatment with degarelix under a clinical study until FE200486 was available on the market or until the study was discontinued.

Study FE200486 CS06A was to provide knowledge of the long-term safety and tolerability of FE200486.

DETAILED DESCRIPTION:
The data include participants from both the main study (FE200486 CS06; NCT00117949) and the extension study FE200486 CS06A.

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet the following inclusion criteria before entry into the study:

* Has given written consent before any study related activity is performed. A study related activity is defined as any procedure that would not have been performed during the normal management of the patient.
* Has had sufficient testosterone suppression (as defined in the withdrawal criteria of FE200486 CS06) for at least 28 days.

Exclusion Criteria:

Any patient meeting any of the following exclusion criteria will not be entered into the study:

* Has been withdrawn from Study FE200486 CS06 due to an adverse event, failure to achieve at least 28 days of testosterone suppression, insufficient prostate-specific antigen (PSA) suppression as defined in Study FE200486 CS06 in the absence of concomitant rise in testosterone level or non-compliance with protocol required procedures.
* Requires hormonal therapy for neoadjuvant purposes.
* Requires treatment with any other drug modifying the testosterone level or function.
* Is considered to be a candidate for curative therapy, i.e., radical prostatectomy or radiotherapy, within 6 months after Visit 1.
* Has a history of severe asthma requiring daily treatment with inhalation steroids, angioedema or anaphylactic reactions.
* Has hypersensitivity towards any component of the investigational product.
* Has had a cancer disease within the last 10 years except for prostate cancer, and surgically removed basocellular or squamous cell carcinoma of the skin.
* Has a clinically significant neurologic, gastrointestinal, renal, hepatic, cardiovascular, psychological, pulmonary, metabolic, endocrine, hematological, dermatological or infectious disorder or any other condition, including excessive alcohol or drug abuse, which may interfere with trial participation or which may affect the conclusion of the study, as judged by the investigator.
* Any clinically significant laboratory abnormalities which, in the judgment of the investigator, would interfere with the patient's participation in this study or evaluation of study results (liver transaminases and bilirubin must be within normal limits).
* Has a mental incapacity or language barrier precluding adequate understanding or co-operation.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2002-10; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (12):
- United States (12):
  - Advanced Urology Medical Center, Anaheim, California
  - South Orange County Medical Research Center, Laguna Woods, California
  - San Bernardino Urological Associates Medical Group, San Bernardino, California
  - Western Clinical Research, Torrance, California
  - Urology Associate PC', Denver, Colorado
  - SW Florida Urological Associates, Fort Myers, Florida
  - Pinellas Urology, Inc., St. Petersburg, Florida
  - Drs. Werner, Murdock & Francis, PA, Greenbelt, Maryland
  - Nevada Urology Associates, Reno, Nevada
  - Urology Specialists of Oklahoma, Inc., Tulsa, Oklahoma
  - Urology Clinics of NorthTexas, PA, Dallas, Texas
  - Urology San Antonio Research, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who responded to degarelix in FE200486 CS06 (NCT00117949) were eligible to enroll into this extension study with the intention of continuing treatment until degarelix became commercially available in the US or until the study was discontinued. Participants received the same dose of degarelix as they received in FE200486 CS06.
Period: Overall Study
Arm/Group | Degarelix 40 mg | Degarelix 80 mg | Degarelix 120 mg | Degarelix 160 mg
Started | 10 | 24 | 24 | 24
Started FE200486 CS06A | 1 | 11 | 16 | 9
Completed | 0 | 4 (Defined as those patients ongoing when the extension study was terminated) | 0 | 3
Not Completed | 10 | 20 | 24 | 21
Not completed — Testosterone >1.0 ng/mL | 9 | 9 | 5 | 9
Not completed — Testosterone 0.5 - 1.0 ng/mL | 1 | 0 | 3 | 2
Not completed — Prostate-specific antigen increase >=25% | 0 | 1 | 5 | 3
Not completed — Other | 0 | 1 | 3 | 1
Not completed — Patient choice | 0 | 0 | 2 | 1
Not completed — Adverse Event | 0 | 2 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 3 | 0
Not completed — PSA decrease <=50% | 0 | 2 | 2 | 4
Not completed — PSA increase >= 10ng/mL | 0 | 1 | 1 | 0
Not completed — Hepatic abnormality | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Degarelix 40 mg | Degarelix 80 mg | Degarelix 120 mg | Degarelix 160 mg | Total
Number analyzed (Participants) | 10 | 24 | 24 | 24 | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2 | 4 | 8
  >=65 years | 9 | 23 | 22 | 20 | 74
Age Continuous [Mean (Standard Deviation); unit: years] | 72.0 (5.72) | 77.5 (6.38) | 75.9 (5.79) | 74.7 (8.37) | 75.6 (6.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 10 | 24 | 24 | 24 | 82
Race/Ethnicity, Customized [Number; unit: participants]
  Black | 2 | 1 | 2 | 1 | 6
  Caucasian | 5 | 23 | 15 | 20 | 63
  Other | 3 | 0 | 7 | 3 | 13
Gleason score [Number; unit: participants] — The Gleason score is a system of grading the aggressiveness of the prostate cancer and how fast it is likely to grow and spread. Scale is 2-10, with low numbers being the least aggressive and 10 being the most aggressive.
  participants
    Unknown | 0 | 1 | 0 | 0 | 1
    2-4 | 1 | 1 | 1 | 0 | 3
    5-6 | 3 | 14 | 12 | 13 | 42
    7-10 | 6 | 8 | 11 | 11 | 36
Stage of prostate cancer [Number; unit: participants] — Prostate cancer stage was classified to describe the extent of cancer. Localized refers to tumors without involvement of lymph nodes or metastasis. Advanced localized can be larger tumors that may involve the lymph nodes but no metastasis. Metastatic are more advanced cancers that are spreading beyond the original tumor.
  participants
    Localized | 5 | 11 | 12 | 10 | 38
    Locally advanced | 0 | 6 | 5 | 5 | 16
    Metastatic | 2 | 4 | 2 | 2 | 10
    Not classifiable | 3 | 3 | 5 | 7 | 18
Body mass index [Mean (Standard Deviation); unit: kilogram per square meter] — Body mass is a measure of body fat based on height and weight.
  kilogram per square meter | 26.7 (5.66) | 26.6 (3.54) | 27.2 (3.15) | 26.6 (3.39) | 26.8 (3.64)
Time since prostate cancer diagnosis [Mean (Standard Deviation); unit: days] — Mean number of days since the participants in each treatment were diagnosed with prostate cancer.
  days | 851 (1077) | 954 (1329) | 1609 (1836) | 1095 (1385) | 1181 (1494)
Weight [Mean (Standard Deviation); unit: kilogram] | 79.0 (11.7) | 81.7 (11.5) | 80.8 (12.8) | 81.4 (14.4) | 81.0 (12.6)

OUTCOME MEASURES:

1. Primary Outcome: Liver Function Tests
Description: The figures present the number of participants who had abnormal (defined as above upper limit of normal range (ULN)) alanine aminotransferase (ALT) levels, aspartate aminotransferase levels, and bilirubin levels plus the number of participants who had ALT increases >3x ULN and ALT increases >3x ULN with concurrently increased bilirubin >1.5 ULN.
Time Frame: 3 years
Population: The data include patients from both the main study (FE200486 CS06) and the extension study FE200486 CS06A.
Measure: Number; unit: participants
Arm/Group | Degarelix 40 mg | Degarelix 80 mg | Degarelix 120 mg | Degarelix 160 mg
Number analyzed (Participants) | 10 | 24 | 24 | 24
participants
  Abnormal alanine aminotransferase (ALAT) | 0 | 4 | 5 | 6
  Abnormal aspartate aminotransferase | 1 | 13 | 18 | 9
  Abnormal bilirubin | 2 | 0 | 4 | 2
  ALAT >3x ULN | 0 | 1 | 0 | 0
  ALAT >3x ULN, bilirubin >1.5x ULN | 0 | 0 | 0 | 0

2. Primary Outcome: Participants With Markedly Abnormal Change in Vital Signs and Body Weight
Description: Vital signs and body weight included incidence of markedly abnormal changes in blood pressure (systolic and diastolic), pulse, and body weight at the end of trial as compared to baseline. The table presents the number of participants in each group with normal baseline and markedly abnormal value post-baseline.
Time Frame: 3 years
Population: These data include patients from the main study (FE200486 CS06) and the extension study (FE200486 CS06A).
Measure: Number; unit: participants
Arm/Group | Degarelix 40 mg | Degarelix 80 mg | Degarelix 120 mg | Degarelix 160 mg
Number analyzed (Participants) | 10 | 24 | 24 | 24
participants
  Diastolic blood pressure <=50 and decrease >=15 | 0 | 1 | 2 | 0
  Diastolic blood pressure >=105 and increase >=15 | 0 | 0 | 0 | 0
  Systolic blood pressure <=90 and decrease >=20 | 0 | 3 | 0 | 1
  Systolic blood pressure >=180 and increase >=20 | 0 | 0 | 1 | 0
  Heart rate <=50 and decrease >=15 | 0 | 1 | 2 | 3
  Heart rate >=120 and increase >=15 | 0 | 0 | 0 | 0
  Body weight decrease of >=7 percent | 0 | 0 | 1 | 0
  Body weight increase of >=7 percent | 0 | 1 | 6 | 1

ADVERSE EVENTS:
Arm/Group | Degarelix 40 mg | Degarelix 80 mg | Degarelix 120 mg | Degarelix 160 mg
Serious Adverse Events (participants affected / at risk) | 0 | 5 | 7 | 2
Other Adverse Events (participants affected / at risk) | 6 | 19 | 21 | 16
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Degarelix 40 mg | Degarelix 80 mg | Degarelix 120 mg | Degarelix 160 mg
Aortic valve incompetence (Cardiac disorders) | 0/10 (0) | 0/24 (0) | 1/24 (1) | 0/24 (0)
Bradycardia (Cardiac disorders) | 0/10 (0) | 0/24 (0) | 1/24 (1) | 0/24 (0)
Cardiac arrest (Cardiac disorders) | 0/10 (0) | 0/24 (0) | 1/24 (1) | 0/24 (0)
Coronary artery disease (Cardiac disorders) | 0/10 (0) | 1/24 (1) | 0/24 (0) | 0/24 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0/10 (0) | 0/24 (0) | 0/24 (0) | 1/24 (1)
Inguinal hernia (Gastrointestinal disorders) | 0/10 (0) | 0/24 (0) | 1/24 (2) | 0/24 (0)
Lobar pneumonia (Infections and infestations) | 0/10 (0) | 0/24 (0) | 1/24 (1) | 0/24 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0/10 (0) | 1/24 (1) | 0/24 (0) | 1/24 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0/10 (0) | 0/24 (0) | 1/24 (1) | 0/24 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0/10 (0) | 0/24 (0) | 1/24 (1) | 0/24 (0)
Blood potassium increased (Investigations) | 0/10 (0) | 1/24 (1) | 0/24 (0) | 0/24 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/10 (0) | 0/24 (0) | 1/24 (1) | 0/24 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/10 (0) | 0/24 (0) | 1/24 (1) | 0/24 (0)
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/10 (0) | 1/24 (1) | 0/24 (0) | 0/24 (0)
Carotid artery stenosis (Nervous system disorders) | 0/10 (0) | 0/24 (0) | 1/24 (1) | 0/24 (0)
Cerebrovascular accident (Nervous system disorders) | 0/10 (0) | 1/24 (1) | 0/24 (0) | 0/24 (0)
Presyncope (Nervous system disorders) | 0/10 (0) | 0/24 (0) | 1/24 (1) | 0/24 (0)
Haematuria (Renal and urinary disorders) | 0/10 (0) | 1/24 (1) | 0/24 (0) | 0/24 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0/10 (0) | 0/24 (0) | 1/24 (1) | 0/24 (0)
Chest pain (General disorders) | 0/10 (0) | 1/24 (1) | 0/24 (0) | 0/24 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Degarelix 40 mg | Degarelix 80 mg | Degarelix 120 mg | Degarelix 160 mg
Anaemia (Blood and lymphatic system disorders) | 0/10 (0) | 2/24 (2) | 5/24 (8) | 0/24 (0)
Angina pectoris (Cardiac disorders) | 0/10 (0) | 2/24 (2) | 1/24 (1) | 0/24 (0)
Constipation (Gastrointestinal disorders) | 0/10 (0) | 4/24 (4) | 2/24 (2) | 2/24 (3)
Diarrhoea (Gastrointestinal disorders) | 0/10 (0) | 2/24 (2) | 4/24 (4) | 0/24 (0)
Inguinal hernia (Gastrointestinal disorders) | 0/10 (0) | 3/24 (4) | 1/24 (1) | 0/24 (0)
Dyspepsia (Gastrointestinal disorders) | 0/10 (0) | 1/24 (1) | 2/24 (2) | 1/24 (2)
Oedema peripheral (General disorders) | 0/10 (0) | 1/24 (1) | 3/24 (4) | 0/24 (0)
Fatigue (General disorders) | 1/10 (1) | 3/24 (3) | 1/24 (1) | 3/24 (4)
Injection site pruritus (General disorders) | 0/10 (0) | 4/24 (4) | 2/24 (2) | 0/24 (0)
Injection site pain (General disorders) | 0/10 (0) | 3/24 (4) | 3/24 (5) | 1/24 (1)
Asthenia (General disorders) | 0/10 (0) | 2/24 (2) | 1/24 (1) | 0/24 (0)
Chest pain (General disorders) | 0/10 (0) | 3/24 (7) | 0/24 (0) | 0/24 (0)
Seasonal allergy (Immune system disorders) | 0/10 (0) | 0/24 (0) | 3/24 (3) | 0/24 (0)
Nasopharyngitis (Infections and infestations) | 0/10 (0) | 3/24 (3) | 3/24 (4) | 3/24 (3)
Urinary tract infection (Infections and infestations) | 0/10 (0) | 3/24 (8) | 1/24 (1) | 1/24 (2)
Influenza (Infections and infestations) | 0/10 (0) | 2/24 (2) | 2/24 (2) | 0/24 (0)
Pharyngitis (Infections and infestations) | 0/10 (0) | 2/24 (2) | 0/24 (0) | 0/24 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0/10 (0) | 3/24 (4) | 0/24 (0) | 0/24 (0)
Injury (Injury, poisoning and procedural complications) | 0/10 (0) | 2/24 (2) | 0/24 (0) | 0/24 (0)
Fall (Injury, poisoning and procedural complications) | 0/10 (0) | 2/24 (2) | 0/24 (0) | 0/24 (0)
Weight increased (Investigations) | 0/10 (0) | 1/24 (1) | 2/24 (2) | 0/24 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0/10 (0) | 2/24 (2) | 0/24 (0) | 0/24 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0/10 (0) | 0/24 (0) | 2/24 (2) | 0/24 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0/10 (0) | 2/24 (3) | 1/24 (1) | 1/24 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1/10 (1) | 1/24 (1) | 0/24 (0) | 1/24 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1/10 (1) | 0/24 (0) | 0/24 (0) | 1/24 (1)
Dizziness (Nervous system disorders) | 1/10 (1) | 3/24 (4) | 3/24 (3) | 1/24 (1)
Headache (Nervous system disorders) | 1/10 (1) | 3/24 (3) | 3/24 (3) | 0/24 (0)
Sciatica (Nervous system disorders) | 0/10 (0) | 2/24 (3) | 0/24 (0) | 0/24 (0)
Dysuria (Renal and urinary disorders) | 0/10 (0) | 3/24 (5) | 1/24 (1) | 2/24 (2)
Urinary retention (Renal and urinary disorders) | 0/10 (0) | 2/24 (2) | 1/24 (1) | 1/24 (1)
Gynaecomastia (Reproductive system and breast disorders) | 0/10 (0) | 4/24 (4) | 1/24 (1) | 1/24 (1)
Testicular atrophy (Reproductive system and breast disorders) | 0/10 (0) | 2/24 (2) | 1/24 (1) | 1/24 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0/10 (0) | 2/24 (2) | 2/24 (2) | 1/24 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0/10 (0) | 2/24 (3) | 1/24 (1) | 0/24 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0/10 (0) | 2/24 (4) | 0/24 (0) | 0/24 (0)
Hot flush (Vascular disorders) | 2/10 (2) | 14/24 (16) | 6/24 (8) | 5/24 (5)
Hypertension (Vascular disorders) | 0/10 (0) | 0/24 (0) | 4/24 (4) | 0/24 (0)
Diabetic retinopathy (Eye disorders) | 1/10 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0)
Haemorrhoids (Gastrointestinal disorders) | 0/10 (0) | 0/24 (0) | 2/24 (2) | 0/24 (0)
Alanine aminotransferase increased (Investigations) | 0/10 (0) | 2/24 (2) | 0/24 (0) | 0/24 (0)
Aspartate aminotransferase increased (Investigations) | 0/10 (0) | 2/24 (2) | 0/24 (0) | 0/24 (0)
Breath sounds abnormal (Investigations) | 1/10 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0)
Libido decreased (Psychiatric disorders) | 0/10 (0) | 1/24 (1) | 2/24 (3) | 3/24 (4)
Urine flow decreased (Renal and urinary disorders) | 1/10 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript.